CLINICAL TRIAL: NCT05367830
Title: A Convergent Parallel Mixed-methods Feasibility Study of the Bone@BC App Version 3.0 to Investigate Feasibility and Satisfaction
Brief Title: A Feasibility Study of the Bone@BC App Version 3.0
Acronym: Believe@BC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Peter Schwarz, Professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2
Record Dates: First submitted 2022-04-19; First posted 2022-05-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the bone@bc app (Experimental): Intervention group patients with breast cancer using the app Bone@BC
  Interventions: Behavioral: the Bone@BC app

INTERVENTIONS:
Behavioral: the Bone@BC app — The bone@BC app is a diary for patients with breast cancer that they can use if they want to.

SUMMARY:
Introduction Due to improvements in diagnostics and treatments, the 5-year survival for patients with breast cancer is 80-90% after initial diagnosis. During treatments, patients typically have consultations weekly and then gradually reduce to annual visits. During this transition from hospital-based care to health self-management, the breast cancer survivors are encouraged to e.g. exercise because of accumulating evidence for the efficacy of exercise training in cancer survivorship, and in the majority of cases, adhere to endocrine treatments to reduce the risk of breast cancer recurrence.

Design and methods The study is a one-arm convergent parallel mixed-methods feasibility intervention study. The quantitative data will be the use of the Bone@bc app (intervention) and questionnaires (n=50) and the Qualitative data will be semi-structured interviews (n= 15 - 20)

DETAILED DESCRIPTION:
AIM The aim is to investigate the feasibility and user satisfaction of an app Bone@BC version 3.0 and if the app Bone@BC can enhance self-efficacy and investigate user statistics and traffic in the app Bone@BC by using a convergent parallel Mixed-Methods design.

Recruitment and procedure For the quantitative data, the recruitment will follow a consecutive sampling strategy, the follow-up group with the electronic patient-reported outcome (ePRO) and systematic consultations (n= 50) will be recruited from the Endocrinology Out-Clinic at Rigshospitalet, Denmark. For the qualitative data, the participants will be recruited from the group participating in the quantitative data following a nested sampling. The patients will be recruited by the principal investigator Trine Lund-Jacobsen (TLJ), or clinical physicians from the Department of Endocrinology, Rigshospitalet, Denmark. The identification of patients will be given to the principal investigator (TLJ) in case the patients are accepted to be contacted for further written and oral information about the project, letter for the subject's rights is handed out and then be provided for obtaining written consent from the patient. The patients who regret or refuse to give consent to participate in the study will be registered and we will note the reason why the patients refuse or regret participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Age 50-70 years
* Danish speaking
* Diagnosed with EBC, stage I-III
* Eligible to receive (neo-) adjuvant chemotherapy or adjuvant treatments
* Access to an E-mail address
* Access to smart mobile electronic devices connected to the internet
* Willingness to have the app installed on the smart mobile electronic devices
* Ability to work with the app

Exclusion Criteria:

* Prior malignancy
* Pre-existing type 2 diabetes or other metabolic diseases
* Withdrawn or not given a consent form

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
The System Usability Scale (SUS) | Week 12
  a self-administrated questionnaire with 10 items with five response options for respondents; from Strongly agree to Strongly disagree. A SUS score above a 68 would be considered above average and anything below 68 is below average.
Feasibility parameters as adherence, acceptability, response rate, representativeness, recruitment rate, and satisfaction | Week 12
  Semi-structured interviews
Bone@BC app | From baseline and to week 12
  Patient-reported outcome(s) from the app on the questions provided daily on Health-Related Quality of Life, late side-effects, symptoms and concerns perspectives, and level of Physical Activity in the app Bone@BC). The daily questions will be from the Eortc Library and will be analysed in percentages.

SECONDARY OUTCOMES:
Changes in symptoms of depression and anxiety measured by Hospital Anxiety and Depression Scale | baseline (0 months) and week 12
  The Hospital Anxiety and Depression scale is a 14-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Changes in Quality of life measured by the European Organization for Research and Treatment of Cancer Quality of Life | baseline (0 months) and week 12
  Health-related quality of life scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Changes in self-efficacy measured by Self-efficacy for managing chronic disease 6-item scale (SES6G) | Week 4, week 8 end week 12
  The Self-efficacy for managing chronic disease 6 item scale is a 6 item scale. Scoring for each item ranges from zero to ten. A high scale score represents a high self-efficacy.
Changes in patient empowerment measured by The Health Education Impact Questionnaire. | baseline (0 months) and week 12
  he Health Education Impact Questionnaire i a 42 items questionnaire with a 4 point response scale (strongly disagree, disagree, agree and strongly agree). Higher values in the Health Education Impact Questionnaire scales indicate better status, except for Emotional distress, where higher values indicate higher distress.
Changes in in app user measured by Open source web analytics application Matomo Analytics | week 4, week 8 and week 12
  In-app user analytics will be collected to track user behavior such as the number of app sessions the user have measured by numbers (quantity).
  Length of app sessions measured by time (hours and sec.). Frequency of use measured in numbers (quantity). Data on when the app was first opened measured as the specific site. Geographic place measured as country. How many pages the users use measured as numbers (quantity). How long time the users spend on the pages measured as time (hours and sec.). Bounce rate measured as numbers (quantity). Returning for the first time measured as numbers (quantity).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schwarz, Principal Investigator — Rigshospitalet, Denmark

REFERENCES:
- [Derived] Lund-Jacobsen T, Schwarz P, Martino G, Pappot H, Piil K. Development of an App for Symptom Management in Women With Breast Cancer Receiving Maintenance Aromatase Inhibitors: Protocol for a Mixed Methods Feasibility Study. JMIR Res Protoc. 2024 Feb 15;13:e49549. doi: 10.2196/49549. PMID 38358787
- [Derived] Lund-Jacobsen T, Bentsen L, Schwarz P, Knop AS, Pappot H, Piil K. Aromatase Inhibitor-Related Symptoms Reported by Postmenopausal Women with Nonmetastatic, Estrogen Receptor-Positive Breast Cancer: A Systematic Review. Semin Oncol Nurs. 2023 Oct;39(5):151487. doi: 10.1016/j.soncn.2023.151487. Epub 2023 Aug 21. PMID 37612223